CLINICAL TRIAL: NCT06157047
Title: Evaluation of the Crestal Bone Expansion Obtained With the Magnetic Mallet® During the Preparation of the Implant Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paolo Pesce (Other)
Responsible Party: Sponsor-Investigator, Paolo Pesce, Prof, Universita degli Studi di Genova
Organization: Universita degli Studi di Genova (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Mallet
Record Dates: First submitted 2023-11-13; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients included (Experimental): Patients' recruitment was guided by their actual need to solve edentulism through the use of implant therapy. The diagnosis was made clinically and radiographically.
  Interventions: Procedure: Crestal Bone Expansion obtained with the Magnetic Mallet®

INTERVENTIONS:
Procedure: Crestal Bone Expansion obtained with the Magnetic Mallet® — A magnetodynamic instrument (Magnetic Mallet®, Metaergonomica, Turbigo, Italy) has been used to perform a horizontal bone expansion in edentulous sites that need to be rehabilitated with a dental implant.

SUMMARY:
The purpose of the study is to evaluate the use of a magnetodynamic instrument (Magnetic Mallet®, Metaergonomica, Turbigo, Italy) to perform a horizontal bone expansion in edentulous sites that need to be rehabilitated with a dental implant.

DETAILED DESCRIPTION:
From October 2019 to May 2022, a sample of 15 patients, 11 men and 4 women, age between 39 and 78 years, was analyzed. A total of 18 conical-shaped implants with a diameter of 3.80 mm and a length between 10 and 11.5 mm were inserted in the maxillary region in the area between the lateral incisor and the first upper molar. The patients were treated by two different surgeons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxillary mono-edentulism between the lateral incisor and the first upper molar with a bone crest measuring between 4-6 mm;
* Insertion of conical implants with dimensions 3.80 x > 10 mm;
* Correct occlusal relationships between upper and lower jaw;
* Patients willing to cooperate and follow the instructions given by the clinicians.

Exclusion Criteria:

* Smokers > 15 cigarettes per day;
* Patients with systemic diseases;
* Irradiation to the head/neck region within 12 months prior to surgery;
* Pregnancy or breastfeeding;
* Poor oral hygiene and lack of motivation to return for checkups;
* Edentulous area for less than 1 year;
* Edentulousness of the lower jaw.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
bone thickness at T0 | Before the surgery
  Thickness of the bone before the surgery measured with cbct and a parodontal probe
bone thickness at T1 | Immediately after the implant site preparation
  Thickness of the bone after the use of Magnetic Mallet measured with a parodontal probe
bone thickness at T2 | Immediately after the implant insertion
  Thickness of the bone after implant insertion measured with a parodontal probe

SECONDARY OUTCOMES:
bone thickness at T3 | 3 months
  Thickness of the bone after 3 months from implant insertion measured with a cbct

CONTACTS AND LOCATIONS:
Locations (1):
- PAD 4 ospedale san martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: No